CLINICAL TRIAL: NCT02430285
Title: Early Endoscopic Ultrasound (EUS) in Acute Biliary Pancreatitis: a Prospective Pilot Study
Brief Title: Early EUS in Acute Biliary Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Chief of Clinical Research, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EARLY-EUS
Record Dates: First submitted 2015-04-07; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Acute Biliary Pancreatitis
Keywords: biliary stone; cholelithiasis; pancreatitis; EUS; ERCP; early; choledocholithiasis
MeSH Terms: conditions — Cholecystolithiasis; Cholelithiasis; Pancreatitis; Choledocholithiasis | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic Ultrasound (Other): All consecutive patients entering the emergency department due to acute abdominal pain and showing biochemical and/or radiological findings consistent with possible acute biliary pancreatitis, undergo Endoscopic Ultrasound with linear array Olympus 180 series echoendoscopes (Olympus Europa Holding, Hamburg, Germany).
  Interventions: Procedure: Endoscopic Ultrasound; Device: Olympus 180 series echoendoscope

INTERVENTIONS:
Procedure: Endoscopic Ultrasound — Endoscopic Ultrasound
  Other Names: Olympus 180 series(Olympus Europa Holding, Hamburg, Germany)
Device: Olympus 180 series echoendoscope

SUMMARY:
Acute biliary pancreatitis (ABP) is a potentially life-threatening condition caused by common bile duct (CBD) stones or sludge, which requires prompt diagnosis and treatment by endoscopic removal of the material. Accurate detection of CBD stones is warranted to select patients for early therapeutic endoscopic retrograde cholangiopancreatography (ERCP).

In clinical practice the decision to perform an ERCP is often based on biochemical and radiological criteria despite they already have been shown to be unreliable predictors of CBD stone presence.

Endoscopic ultrasound (EUS) is not currently a worldwide standard diagnostic procedure early in the course of acute biliary pancreatitis, but it has been shown to be accurate, safe and cost effective in diagnosing biliary obstructions compared with magnetic resonance cholangiopancreatography (MRCP) and ERCP and therefore in preventing unnecessary ERCP and its related complications.

The investigators aim to investigate the clinical usefulness of early EUS in the management of ABP.

All consecutive patients entering the emergency department due to acute abdominal pain and showing biochemical and/or radiological findings consistent with possible ABP will be prospectively enrolled. Patients will be classified as having a low, moderate, or high probability of CBD stones, according to established risk stratification. All enrolled patients will undergo EUS within 48 h of their admission. ERCP will be performed immediately after EUS only in those cases with proven CBD stones or sludge.

The following parameters will be investigated: (1) clinical: age, sex, fever; (2) radiological: dilated CBD, (3) biochemical: bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase (gGT), alkaline phosphatase (ALP), amylase, lipases, C-reactive protein (CRP). Association between presence of CBD stone at EUS and the individual predictors were assessed by univariate logistic regression. Predictors significantly associated with CBD stones (p<0.05) will enter in a multivariate logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients entering the emergency department for possible acute biliary pancreatitis

Exclusion Criteria:

* gastrectomy
* patient in whom the cause of biliary obstruction was already identified by US

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Reliability of early EUS | Twenty-four hours
  Accuracy of EUS in detecting CBD stones (percentage of detection of choledocholithiasis with an early EUS approach in all patients with ABP)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Anderloni, MD, PhD, Principal Investigator — Digestive Endoscopy Unit, Division of Gastroenterology, Humanitas Research Hospital, Rozzano, Milan, 20089, Italy
Locations (1):
- Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milan, Italy, Italy

REFERENCES:
- [Background] Fabbri C, Polifemo AM, Luigiano C, Cennamo V, Fuccio L, Billi P, Maimone A, Ghersi S, Macchia S, Mwangemi C, Consolo P, Zirilli A, Eusebi LH, D'Imperio N. Single session versus separate session endoscopic ultrasonography plus endoscopic retrograde cholangiography in patients with low to moderate risk for choledocholithiasis. J Gastroenterol Hepatol. 2009 Jun;24(6):1107-12. doi: 10.1111/j.1440-1746.2009.05828.x. PMID 19638088
- [Background] ASGE Standards of Practice Committee; Maple JT, Ben-Menachem T, Anderson MA, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Strohmeyer L, Dominitz JA. The role of endoscopy in the evaluation of suspected choledocholithiasis. Gastrointest Endosc. 2010 Jan;71(1):1-9. doi: 10.1016/j.gie.2009.09.041. No abstract available. PMID 20105473
- [Background] De Lisi S, Leandro G, Buscarini E. Endoscopic ultrasonography versus endoscopic retrograde cholangiopancreatography in acute biliary pancreatitis: a systematic review. Eur J Gastroenterol Hepatol. 2011 May;23(5):367-74. doi: 10.1097/MEG.0b013e3283460129. PMID 21487299
- [Derived] Anderloni A, Galeazzi M, Ballare M, Pagliarulo M, Orsello M, Del Piano M, Repici A. Early endoscopic ultrasonography in acute biliary pancreatitis: A prospective pilot study. World J Gastroenterol. 2015 Sep 28;21(36):10427-34. doi: 10.3748/wjg.v21.i36.10427. PMID 26420969